CLINICAL TRIAL: NCT00645034
Title: A Double-blind, Placebo-controlled, Randomized, 2-way Crossover Study to Investigate the Hemodynamic Effects of a Single Dose of Sildenafil (100mg) in Subjects With Benign Prostatic Hyperplasia Being Treated With Doxazosin
Brief Title: A Study to Investigate the Effects on Blood Pressure and Pulse Rate of a Single 100mg Dose of Sildenafil in Patients With Benign Prostatic Hyperplasia Who Are Being Treated With Doxazosin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: A1481163
Record Dates: First submitted 2008-03-20; First posted 2008-03-27 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: sildenafil
- Arm 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — placebo by mouth as a single dose
  Arms: Arm 2
Drug: sildenafil — sildenafil 100 mg by mouth as a single dose
  Arms: Arm 1

SUMMARY:
To investigate the effects of a single dose of sildenafil (100 mg) or placebo on blood pressure and pulse rate in subjects taking doxazosin for benign prostatic hyperplasia (BPH). To investigate the pharmacokinetics of doxazosin when co-administered with sildenafil 100 mg, and to investigate the safety and toleration of sildenafil 100 mg when co-administered with doxazosin.

ELIGIBILITY:
Inclusion Criteria:

* patients who weighed between 132 and 220 lb (60 and 100 kg) with benign prostatic hyperplasia (BPH)
* a total PSA (prostate specific antigen) measurement of less than or equal to 10 µg/L within the 12 months prior to screening, were currently on doxazosin treatment for BPH, had been treated with doxazosin for a minimum of 2 months prior to first dose of study medication, and had received a minimum of 4 mg doxazosin once daily (from doxazosin supplied for this study) for 2 weeks prior to the first dose of study medication.

Exclusion Criteria:

* subjects with a recent history (i.e. within 6 months prior to screening) of stroke or myocardial infarction
* subjects with severe cardiovascular disorders such as unstable angina or severe congestive heart failure
* subjects with known hereditary degenerative retinal disorders, such as retinitis pigmentosa
* subjects with a supine systolic/diastolic blood pressure of >170/100 mmHg or <100/60 mmHg either at screening or at the pre-dose measurements
* subjects receiving any other antihypertensive therapy other than doxazosin in the 3 weeks prior to the first dose of study medication.

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-11; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic parameters of blood pressure and pulse rate | immediately predose, 15, 30, and 45 minutes and 1, 1.5, 2, 2.5, 3, 4, 6, and 8 hours postdose

SECONDARY OUTCOMES:
Blood samples for doxazosin pharmacokinetic parameters | time 0 (pre-dose), and at 1, 2, 3, 4, 6, and 8 hours post-dose
Safety and toleration of simultaneously co-administering sildenafil and doxazosin. | continuous

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Laguna Woods, California
  - Pfizer Investigational Site, Newport Beach, California